CLINICAL TRIAL: NCT02811978
Title: A Phase 3, Randomized, Open-label Study of Subcutaneous and Intravenous VELCADE in Combination With Dexamethasone in Chinese Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Subcutaneous and Intravenous Velcade in Combination With Dexamethasone in Chinese Subjects With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108175; 26866138MMY3037 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-05-26; First posted 2016-06-23 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : Intravenous Bortezomib plus Dexamethasone (Experimental): Participants will receive a 1.3 milligram per square meter per dose (mg/m^2) bortezomib intravenously on Days 1, 4, 8, and 11 of a 3 week cycle. Participants will receive Dexamethasone at a dose of 20 mg oral (PO) on the day of and the day after bortezomib dosing (Days 1, 2, 4, 5, 8, 9, 11, and 12 of each cycle).
  Interventions: Drug: Bortezomib; Drug: Dexamethasone
- Group 2 : Subcutaneous Bortezomib plus Dexamethasone (Experimental): Participants will receive a 1.3 milligram per square meter per dose (mg/m^2) bortezomib subcutaneously on Days 1, 4, 8, and 11 of a 3 week cycle. Participants will receive Dexamethasone at a dose of 20 mg oral (PO) on the day of and the day after bortezomib dosing (Days 1, 2, 4, 5, 8, 9, 11, and 12 of each cycle).
  Interventions: Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Participants will receive 1.3 mg/m^2 bortezomib on Days 1, 4, 8, and 11 of a 3 week cycle.
  Other Names: Velcade; JNJ-26866138-AAA
Drug: Dexamethasone — Participants will receive Dexamethasone at a dose of 20 mg PO on the day of and the day after bortezomib dosing (Days 1, 2, 4, 5, 8, 9, 11, and 12 of each cycle).

SUMMARY:
The purpose of this phase 3 study is to determine if subcutaneous velcade is non-inferior to intravenous velcade when administered in combination with low-dose dexamethasone in chinese refractory or relapsed multiple myeloma (r/rMM) patients. The study will assess the overall response rate after 4 cycles of velcade and dexamethasone administration.

ELIGIBILITY:
Inclusion Criteria:

* Have received at least 1 and no more than 3 prior lines of therapy for multiple myeloma
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* The toxicities resulting from previous therapy must be resolved or stabilized to less than or equal (<=)Grade 1 prior to drug administration
* A woman of childbearing potential must have a negative highly sensitive serum (human chorionic gonadotropin [hCG]) or urine pregnancy tests at screening within 14 days prior to Cycle 1 Day 1
* Have documented evidence of progressive disease/disease progression based on investigator's determination of response by the International Myeloma Working Group (IMWG) criteria on or after their last regimen

Exclusion Criteria:

* Received antimyeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before the date of randomization. The only exception is emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 milligram per day (mg/day) for a maximum of 4 days) before treatment.
* Received autologous stem cell transplant (ASCT) within 12 weeks before the date of randomization, or the participant has previously received an allogenic stem cell transplant (regardless of timing)
* Plans to undergo a stem cell transplant prior to progression of disease on this study, that is, these participants should not be enrolled in order to reduce disease burden prior to transplant
* Is known to be infected with human immunodeficiency virus (HIV) or active infection with hepatitis B or hepatitis C
* Had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or clinically significant conduction system abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate After 4 Cycles of Velcade Treatment | 12 weeks (after 4 cycles; each cycle is of 3 weeks)
  ORR defined as the proportion of participants who achieve either complete response [CR], very good partial response [VGPR], or partial response [PR], according to the International Myeloma Working Group (IMWG) criteria. Participants with CR, VGPR, or PR that is unconfirmed in Cycle 4 but confirmed in the next response assessment will be included as CR, VGPR or PR, respectively.

SECONDARY OUTCOMES:
Complete Response (CR) and Very Good Partial Response (VGPR) after 4 cycles | 12 weeks (after 4 cycles; each cycle is of 3 weeks)
  CR and VGPR defined as the proportion of participants who achieve either complete response [CR] or very good partial response [VGPR], according to the IMWG criteria, after 4 cycles of Velcade treatment. Participants with CR or VGPR that is unconfirmed in Cycle 4 but further confirmed in the next response assessment will be included.
Overall Response Rate (ORR) after 8 cycles | 24 weeks (after 8 cycle; each cycle is of 3 weeks)
  ORR is defined as the proportion of participants who achieve either CR, VGPR, or PR according to the IMWG criteria, after 8 cycles of Vd treatment. Participants with CR, VGPR or PR that is unconfirmed in Cycle 8 but further confirmed in the next response assessment will be included.
Progression-Free Survival (PFS) | Maximum up to 4 years 7 months
  PFS is defined as the time from the date of randomization to the date of first documented progressive disease/disease progression (PD), or death due to any cause, whichever occurs earlier. Participants who have not progressed and are alive on the cut-off date for analysis will be censored at the date of the last clinical assessment of response.
One-year survival rate | 1 year after last patient randomization
  One-year survival rate is defined as survival rate at 1 year after randomization. If a participant is alive or the vital status is unknown, then data will be censored at the date that the participant is last known to be alive.
Time to response | Maximum up to 4 years 7 months
  Time to response is defined as the time from the date of randomization to the date of the first documentation of a confirmed CR, VGPR, or PR. Participants without response (CR/VGPR/PR) will be censored either at PD or at the last clinical assessment of response.
Time to progression (TTP) | Maximum up to 4 years 7 months
  Time to progression is defined as the time from the date of randomization to the date of first documentation of PD. Participants who have not progressed will be censored at the date of the last clinical assessment of response.
Duration of response (DOR) | Maximum up to 4 years 7 months
  Duration of response is defined as the time from the date of first documentation of a confirmed CR, VGPR, or PR (overall cycles) to the date of first documented PD. Responders without PD will be censored at the date of the last clinical assessment of response.
Time to best response | Maximum up to 4 years 7 months
  Time to best response is defined as the time from the date of randomization to the date of the first evaluation of the overall best response (CR/VGPR/PR) to treatment. Participants without response (CR/VGPR/PR) will be censored either at PD or at the last clinical assessment of response.
Maximum Observed Plasma Concentration (Cmax) | Cycle 1 of Day 1, Day 11 to Day 14
  Drug concentration vs. time profile following the 4th dose in Cycle 1 and derived Pharmacokinetic (PK) parameter Cmax will be assessed. Cmax is the observed maximum plasma concentration, taken directly from the plasma concentration-time profile.
Area Under the Plasma ConcentrationTime Curve From Time 0 to Last Observed Quantifiable Concentration AUC [0-last] | Cycle 1 of Day 1, Day 11 to Day 14
  Drug concentration vs. time profile following the 4th dose in Cycle 1 and derived Pharmacokinetic (PK) parameter AUC [0-last] will be assessed. AUC [0-last] is the area under the plasma-concentration versus time curve from time 0 to the time of last quantifiable time point, calculated by linear trapezoidal summation.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Cycle 1 of Day 1, Day 11 to Day 14
  Drug concentration vs. time profile following the 4th dose in Cycle 1 and derived Pharmacokinetic (PK) parameter Tmax will be assessed. Tmax is the time when Cmax is observed, taken directly from the plasma concentration-time profile.
Number of Participants with Treatment-Related Adverse Events and Serious Treatment-Related Adverse Events | Maximum up to 4 years 7 months
  Number of Participants with adverse events will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0.3 and also vital signs, clinical laboratory tests, local injection site tolerability, and electrocardiograms (ECGs) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- China (10):
  - Beijing
  - Chengdu
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Nanjing
  - Shanghai
  - Suzhou
  - Tianjin
  - Wuhan

REFERENCES:
- See also: A Phase 3, Randomized, Open-label Study of Subcutaneous and Intravenous VELCADE® in Combination with Dexamethasone in Chinese Subjects with Relapsed or Refractory Multiple Myeloma — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108175&attachmentIdentifier=77e89ae3-7f6b-4eb6-8499-925c2be8f4d6&fileName=CR108175_CSR_Synopsis.pdf&versionIdentifier=